CLINICAL TRIAL: NCT07351305
Title: Non-Trauma Intervention to Treat Posttraumatic Stress Disorder (PTSD) for Veterans and Service Members Suffering From a Traumatic Brain Injury (TBI)
Brief Title: Non-Trauma Intervention to Treat PTSD for Veterans and Service Members Suffering From a TBI
Acronym: T3 for PTSD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Cindy McGeary, Professor, The University of Texas Health Science Center at San Antonio
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00001920; HT94252411015 (Other: Department of Defense Traumatic Brain Injury and Psychological Health Research Program)
Record Dates: First submitted 2026-01-09; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: mTBI - Mild Traumatic Brain Injury; PTSD; Post Traumatic Stress Disorder
Keywords: Non-trauma intervention; Veterans; Service Members
MeSH Terms: conditions — Brain Concussion; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: This study is a single group pilot test
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Active duty service members and veterans seeking clinical care for mTBI (Experimental): Male and female active duty service members and veterans at least 18 years of age who are seeking clinical care for mild Traumatic Brain Injury (TBI) symptoms at the Intrepid Spirit Center located on Fort Hood who also have a co-occurring diagnosis of PTSD
  Interventions: Behavioral: Non-Trauma Treatment for mTBI and PTSD

INTERVENTIONS:
Behavioral: Non-Trauma Treatment for mTBI and PTSD — The treatment includes 8 sessions with each session lasting approximately 60 minutes. Sessions will cover relaxation training, identifying stress, stress management, and problem solving.
  Other Names: T3 PTSD

SUMMARY:
The investigators want to test a treatment for posttraumatic stress disorder (PTSD) especially designed for military veterans and service members with mild traumatic brain injuries (TBI) and PTSD. The treatment will include individual psychotherapy sessions to manage PTSD.

DETAILED DESCRIPTION:
The objective of this study is to test a non-trauma intervention for PTSD tailored to military veterans and service members with mTBI called Non-Trauma Treatment for TBI and comorbid PTSD (T3 PTSD).

Aim1:

Conduct a pilot study of the non-trauma intervention for comorbid mTBI and PTSD in a sample of n = 20 veterans and service members seeking treatment at Fort Hood, Texas.

Aim2:

Establish the acceptability and feasibility of the non-trauma intervention in service members and veterans.

ELIGIBILITY:
Inclusion Criteria:

1. Ability of participant to understand and the willingness to sign a written informed consent document based on interviewer assessment and clinical judgement.
2. Any veteran or active duty service member (age 18 or above) diagnosed with mTBI as determined by the Ohio State University Brain Injury Identification Method
3. Participant meets diagnostic criteria for PTSD based on Clinician-Administered PTSD Scale (CAPS-5) interview with at least moderate severity (as described by the National Center for PTSD) which includes at least one Criterion B symptom, one Criterion C symptom, two Criterion D symptoms, and two Criterion E symptoms as well as meeting Criterions F and G.
4. Participant is stable on medications at baseline assessment (i.e., no changes in medication prescriptions in the past 4 weeks).
5. Ability to read, write, and speak English based on interviewer assessment and clinical judgement.

Exclusion Criteria:

1. Participant is actively engaged in a behavioral intervention primarily targeting PTSD.
2. Participant has a psychiatric problem that warrants immediate treatment as indicated in the electronic health record, flagged during testing, or confirmed by a clinician through screening or review of clinical notes.
3. Participant demonstrates significant cognitive impairment that could impact treatment adherence/benefit based on interviewer assessment and clinical judgement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
PTSD Checklist-DSM-5 (PCL-5) | Baseline to 6 months post treatment (approximately 8 months)
  The PCL-5 is a 20-item self-report measure designed to assess PTSD symptoms as defined by the DSM-5. The scoring involves summing the responses to 20 items (0 to 80) with higher scores indicating more severe PTSD.

SECONDARY OUTCOMES:
Credibility and Expectancy Questionnaire | Baseline to 2 weeks post treatment (approximately 10 weeks)
  A 6-item measure that was designed to assess treatment expectancy and rationale credibility for use in clinical outcomes studies. The measure is scored on an 8-point scale with higher scores indicating higher credibility and expectancy.
Clinician Administered PTSD Scale for the Diagnostic and Statistical Manual of Mental Disorders Version 5 (DSM-5) | Baseline to 6 months post treatment (approximately 8 months)
  The CAPS-5 contains 20-items measuring PTSD symptoms, scored on a 5-point scale with scores ranging from 0-80. Higher scores indicate greater PTSD severity.
Generalized Anxiety Disorder-7 (GAD-7) | Baseline to 6 months post treatment (approximately 8 months)
  This 7-item measure asks participants to rate the frequency with which they have been bothered by anxiety symptoms within the past 2 weeks. Scores range from 0=not at all to 3=nearly every day, with totals from 0-21, with a higher score indicating greater anxiety.
Patient Global Impressions (PGI) Scale | 2 weeks post treatment to 6 months post treatment
  A 2-item survey where each item is scored out of 7. Total score is 0-14, where a lower score indicates less feeling of illness and greater improvement
Alcohol Use Disorders Identification Test (AUDIT) | Baseline to 6 months post treatment (approximately 8 months)
  A self report, 10-item survey with items scored from 0-4. Total scores range from 0-40, with a higher score indication greater alcohol consumption.
Patient Health Questionnaire-9 (PHQ-9) | Baseline to 6 months post treatment (approximately 8 months)
  The PHQ-9 is a widely used and well-validated 9-item instrument for measuring the severity of depressive symptoms. Each item is scored from 0=not at all to 3=nearly every day giving a possible range of score from 0-27. A lower score indicates better health and well-being
Depressive Symptom Index-Suicide Subscale (DSI-SS) | Baseline to 6 months post treatment (approximately 8 months)
  This 4-item self-report measure of suicidal ideation has excellent internal consistency and concurrent validity. Items are scored 0-3, giving a total range of 0-12, with a higher score indicating more severe suicidal ideation.
Insomnia Severity Index (ISI) | Baseline to 6 months post treatment (approximately 8 months)
  A 7 item scale scored from 0-4 for each item. Total scores range from 0-28 with a higher score indicating worse insomnia.
Life Events Checklist-5 (LEC-5) | Baseline to 6 months post treatment (approximately 8 months)
  The LEC-5 includes a list of 16 potentially traumatic life events commonly associated with PTSD symptoms, along with an additional item (17) that allows respondents to describe any other stressful events or experience. For each potentially traumatic life event, respondents rate their experience of that event on a 6-point nominal scale (1 = happened to me, 2 = witnessed it, 3= learned about it, 4 = part of my job, 5 = not sure, and 6 = doesn't apply). Total scores range from 6-102, with a higher score indicating less traumatic events.
Satisfaction with Therapy and Therapist Scale (STTS) | 2 weeks post treatment (approximately 10 weeks after the first treatment)
  A 12-item self-report measure with strong psychometric properties used to assess the patient's satisfaction with the therapy provided and the therapist. Even number items assess satisfaction with therapy and odd number items assess satisfaction with therapist. Scores range between 5-60 with higher scores reflective of greater satisfaction. Items are on a 5-point Likert scale that ranges from 1 = "Strong disagree" to 5 = "Strongly Agree'. Additionally, a 13th item provides an independent assessment of the patient's global improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Cindy McGeary, PhD, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- Carl R Darnall Army Medical Center, Fort Hood, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual Participant data may be shared with the research study team, the IRB, the Department of Defense representatives and state or Federal Government officials where required by law. Only deidentified data will be shared in a peer reviewed journal or in the summary results in ClinicalTrials.gov.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Public data will be shared at the end of the study after the data is analyzed.